CLINICAL TRIAL: NCT01675063
Title: Development of a Minimally Invasive Cardiac Output Monitoring Device for Critically Ill Patients
Brief Title: Minimally Invasive Cardiac Output Monitoring Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Retia Medical (Unknown)
Responsible Party: Principal Investigator, Dr. James M. Blum, Assistant Professor Of Anesthesiology, Director of Critical Care Research, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UM HUM 63973
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Cardiac Event
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Retia Non-Invasive Sensors (Other): Sensors will be placed on the patient and connected to an amplifier that produces a waveform for 8 hours post cardiac surgery.
  Interventions: Device: Retia Non-Invasive Sensors

INTERVENTIONS:
Device: Retia Non-Invasive Sensors — Three adhesive sensor patches (similar to ECG patches) will be placed on the chest and a sensor similar to a pulse oximeter will be placed on the toe. The sensors will be connected to an electrical amplifier that produces a waveform.

SUMMARY:
The overall goal of this collaborative study is to advance the novel "pulse contour analysis" to the point at which it can be incorporated into a real-time device. The specific objective is to establish an auto-calibration algorithm that conveniently yields cardiac output (CO) in units of liters-per-minute. To achieve this objective, the waveforms for analysis and reference pulmonary artery catheter CO measurements will be recorded from critically ill patients and then analyzed off-line at Retia Medical. Successful completion of this study may ultimately help lead to improved outcomes of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the University of Michigan ICU following cardiac surgery with both a pulmonary and radial artery catheter.

Exclusion Criteria:

* Adult patients with mechanical cardiac support including intra-aortic balloon pumps, LVAD, or ECMO, and persistent ventricular arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2012-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Blum, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Retia Non-Invasive Sensors
Started | 77
Completed | 77
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Retia Non-Invasive Sensors
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 49
Age, Continuous [Mean (Full Range); unit: years] | 69 [35 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 46
Region of Enrollment [Number; unit: participants]
  United States | 77

OUTCOME MEASURES:

1. Primary Outcome: Establishment of a Dataset to Create an Algorithm to Measure Cardiac Output
Description: The primary outcome of this work is to establish a dataset that would enable the calculation of a predicted cardiac output using waveform analysis from multiple sensors. The primary outcome of this work is the number of subjects that successfully contributed data.
Time Frame: 8 hours post cardiac surgery
Population: patients had undergone routine cardiac surgery. some patients did not have PA catheters placed and subsequently data was not obtained on cardiac output.
Measure: Count of Participants; unit: Participants
Arm/Group | Retia Non-Invasive Sensors
Number analyzed (Participants) | 77
Participants
  analyzable data obtained | 75
  data flawed and unable to analyze | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Retia Non-Invasive Sensors
Serious Adverse Events (participants affected / at risk) | 0/77
Other Adverse Events (participants affected / at risk) | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is not involved with the ultimate analysis of the data which is to be used for proprietary algorithm development. The PI was engaged with his opinion on algorithm development and review of waveform data.